CLINICAL TRIAL: NCT01715831
Title: A Multicenter, Open-Label, Single-Arm Extension Study to Describe the Safety of Tocilizumab Treatment In Brazilian Patients With DMARDs Refractory Rheumatoid Arthritis Which Completed Studies ML21530 and MA21488 and Presenting an Indication of Maintaining the Tocilizumab Treatment
Brief Title: A Long-term Safety Extension Study of Tocilizumab in Brazilian Participants With Rheumatoid Arthritis (RA) Who Completed the Studies ML21530 and MA21488
Acronym: RITACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28091
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab 8 mg/kg IV infusion every 4 weeks for a total of 104 weeks. The maximum single dose administered to any participant will be of 800 mg of tocilizumab. Participants may also receive disease-modifying anti-rheumatic drugs (DMARDs) in addition to the tocilizumab treatment in any visit, at the investigator discretion, according to the local prescription information and participant's tolerance.
  Interventions: Drug: DMARDs; Drug: Tocilizumab

INTERVENTIONS:
Drug: DMARDs — DMARDs may be added to the tocilizumab treatment in any visit, at the discretion of the investigator, according to the local prescription information and participant's tolerance. Study protocol does not specify any particular DMARD.
Drug: Tocilizumab — Tocilizumab will be administered at 8 mg/kg IV dose every 4 weeks for 104 weeks
  Other Names: RoActemra; Actemra

SUMMARY:
This multicenter, open-label, single-arm extension study will evaluate the long-term safety of tocilizumab (RoActemra/Actemra) in participants with RA. Participants who have completed the MA21488 (NCT00810199) core study and the ML21530 (NCT00754572) study and who could benefit from the study drug, according to the opinion of the investigator, will receive 8 milligrams per kilogram (mg/kg) of intravenous (IV) tocilizumab every 4 weeks. The anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed their last visit in the core studies ML21530 and MA21488 and that might benefit from treatment using the study drug according to the investigator's evaluation
* Absence of an AE or current or recent laboratory finding that would prevent the use of the 8 mg/kg dose of the tocilizumab
* Receiving outpatient treatment
* For women who are not postmenopausal and are not surgically sterile: agreement to use at least one adequate method of contraception

Exclusion Criteria:

* Participants who have prematurely discontinued the core studies ML21530 and MA21488 for any reason
* MA21488 study participants who remained untreated with tocilizumab after it's discontinuation according to the treatment-free remission criteria of MA21488 study
* Immunization with a live/attenuated vaccine since the last administration of the study drug in the core studies ML21530 and ML21488
* Diagnosis after the last visit of the study ML21530 or after the last visit of the study MA21488 of a rheumatic autoimmune disease other than RA, including systemic erythematous lupus (SEL), mixed connective tissue disease (MCTD), scleroderma and polymyositis, or a significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's syndrome). Secondary Sjogren's Syndrome and/or nodulosis with RA are allowed
* Diagnosis after the last visit of the core study ML21530 or of the study MA21488 of an inflammatory joint disease other than RA
* Abnormal laboratory parameters at the baseline
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Evidences of a concomitant, serious and uncontrolled illness
* Known active condition or a history of recurrent infections by bacteria, viruses, fungi, mycobacteria or other agents
* Evidence of an active malignant disease, malignancies diagnosed in the last 10 years or breast cancer diagnosed in the last 20 years
* Uncontrolled disease status, such as asthma or inflammatory bowel disease in which acute crises are usually treated with oral or parenteral corticosteroids
* Current hepatic disease, as determined by the investigator
* Active tuberculosis (TB) requiring treatment in the previous three years. Participants should be screened for latent TB according to local practice guidelines and should not be admitted into the study if latent TB is detected. Participants must not present any evidence of active TB infection at the enrollment. Participants treated for tuberculosis without recurrence in three years are allowed
* History of alcohol, drugs or chemical abuse since the inclusion in the core studies ML21530 and MA21488

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2016-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Brazil (9):
  - Hospital Universitario Cassiano Antonio Moraes - UFES; Reumatologia, Vitória, Espírito Santo
  - Santa Casa de Misericordia de Salvador; Reumatologia, Salvador, Estado de Bahia
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP; Reumatologia, São Paulo, São Paulo
  - Hospital Abreu Sodre - AACD;Reumatologia, São Paulo, São Paulo
  - Hospital Estadual do Servidor Publico; Reumatologia, São Paulo, São Paulo
  - Centro Paulista de Investigacao Clinica - CEPIC, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 4 weeks for a total of 104 weeks. The maximum single dose administered to any participant was 800 mg of tocilizumab. Participants might have also received disease-modifying anti-rheumatic drugs (DMARDs) in addition to the tocilizumab treatment in any visit, at the investigator discretion, according to the local prescription information and participant's tolerance.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 26
Completed | 25
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population included all participants who received at least one dose of tocilizumab during the study.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV infusion every 4 weeks for a total of 104 weeks. The maximum single dose administered to any participant was 800 mg of tocilizumab. Participants might have also received DMARDs in addition to the tocilizumab treatment in any visit, at the investigator discretion, according to the local prescription information and participant's tolerance.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-Serious Adverse Events (NSAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; significant medical event, according to the investigator discretion (e.g., may represent a risk to the participant or may require medical/surgical intervention to prevent one of the outcomes mentioned above).
Time Frame: From Baseline up to approximately 2 years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
participants
  SAEs | 4
  NSAEs | 24

2. Primary Outcome: Number of Participants With AEs Leading to Dose Modification or Study Discontinuation
Time Frame: From Baseline up to approximately 2 years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
participants
  AEs leading to dose modification | 7
  AEs leading to study discontinuation | 1

3. Primary Outcome: Number of Participants With AEs of Special Interest
Description: Adverse events of special interest included following events: Infections (including opportunistic infections); myocardial infarction / acute coronary syndrome; gastrointestinal (GI) perforations and related events; malignancies; anaphylaxis/hypersensitivity reactions; demyelinating disorders; stroke; hemorrhagic events; and hepatic events. Overall number of participants who experienced any of these AEs of special interest was reported.
Time Frame: From Baseline up to approximately 2 years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
participants | 0

4. Secondary Outcome: Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: DAS28 score is a measure of participant's disease activity calculated using tender joint count in 28 joints (TJC28), swollen joint count in 28 joints (SJC28), participant's global assessment of disease activity (general health [GH]) using visual analog scale (VAS), 0 millimeter (mm)=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS, and acute phase response (erythrocyte sedimentation rate [ESR] in millimeters per hour [mm/hr]) for a total possible score of 0 to 10. The score is calculated using the following formula: DAS28 = [0.56 multiplied by (*) square root (√) of TJC28] plus (+) [0.28*√SJC28]+[0.70*the natural logarithm (ln) ESR]+[0.014*GH]. DAS28-ESR score varies from 0 to 10, where higher scores represent greater disease activity.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and follow-up (FU) Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
units on a scale
  Baseline (n=26) | 2.76 (1.19)
  Week 12 (n=24) | 2.23 (0.86)
  Week 24 (n=25) | 2.43 (1.01)
  Week 36 (n=25) | 2.04 (0.85)
  Week 48 (n=21) | 2.32 (1.23)
  Week 56 (n=24) | 1.82 (0.55)
  Week 68 (n=23) | 2.21 (0.84)
  Week 80 (n=24) | 2.06 (0.64)
  Week 92 (n=24) | 2.23 (0.96)
  Week 104 (n=25) | 1.92 (0.93)
  FU Visit 1 (n=13) | 1.70 (1.02)
  FU Visit 2 (n=24) | 3.21 (1.35)

5. Secondary Outcome: Tender Joint Count (TJC)
Description: An assessment of 28 joints was conducted for tenderness. Joints were assessed and classified as tender/not tender by pressure and joint manipulation after a physical examination. Artificial joints, arthrodesis or fused joints were not taken into consideration for tenderness.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
tender joints
  Baseline (n=26) | 2.8 (3.6)
  Week 12 (n=24) | 1.8 (2.3)
  Week 24 (n=25) | 2.0 (3.6)
  Week 36 (n=25) | 1.9 (2.5)
  Week 48 (n=21) | 2.8 (3.8)
  Week 56 (n=24) | 1.1 (1.2)
  Week 68 (n=23) | 2.0 (2.6)
  Week 80 (n=24) | 1.6 (2.0)
  Week 92 (n=24) | 1.5 (1.7)
  Week 104 (n=25) | 1.5 (1.8)
  FU Visit 1 (n=13) | 1.8 (3.7)
  FU Visit 2 (n=24) | 2.8 (4.7)

6. Secondary Outcome: Swollen Joint Count (SJC)
Description: An assessment of 28 joints was conducted for swelling. Joints were assessed and classified as swollen/not swollen by pressure and joint manipulation after a physical examination. Artificial joints, arthrodesis or fused joints were not taken into consideration for swelling.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
swollen joints
  Baseline (n=26) | 1.4 (2.0)
  Week 12 (n=24) | 1.0 (2.0)
  Week 24 (n=25) | 0.6 (1.2)
  Week 36 (n=25) | 0.9 (1.0)
  Week 48 (n=21) | 1.4 (2.5)
  Week 56 (n=24) | 0.8 (1.8)
  Week 68 (n=23) | 0.9 (1.5)
  Week 80 (n=24) | 0.4 (0.8)
  Week 92 (n=24) | 0.8 (1.2)
  Week 104 (n=25) | 0.6 (1.3)
  FU Visit 1 (n=13) | 0.2 (0.4)
  FU Visit 2 (n=24) | 1.5 (2.2)

7. Secondary Outcome: Global Evaluation of Disease Activity by the Participant Using VAS Score
Description: Participant's global assessment of disease activity was measured on a horizontal 0-100 mm VAS, with 0 mm (left end of the line) described as "inactive disease" (free of symptoms and without symptoms of arthritis) and 100 mm (right end of the line) as "disease maximum activity" (maximum activity of arthritis). The participant marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
mm
  Baseline (n=26) | 35.2 (25.3)
  Week 12 (n=26) | 36.4 (26.4)
  Week 24 (n=26) | 38.4 (27.2)
  Week 36 (n=25) | 31.8 (25.0)
  Week 48 (n=23) | 32.8 (28.8)
  Week 56 (n=25) | 30.6 (22.7)
  Week 68 (n=24) | 32.4 (24.6)
  Week 80 (n=24) | 36.1 (26.2)
  Week 92 (n=25) | 36.2 (25.5)
  Week 104 (n=25) | 33.4 (25.2)
  FU Visit 1 (n=15) | 37.1 (28.0)
  FU Visit 2 (n=25) | 42.6 (29.9)

8. Secondary Outcome: Global Evaluation of Disease Activity by the Physician Using VAS Score
Description: Physician global assessment of disease activity was measured on a horizontal 0-100 mm VAS, with 0 mm (left end of the line) described as "inactive disease" (free of symptoms and without symptoms of arthritis) and 100 mm (right end of the line) as "disease maximum activity" (maximum activity of arthritis). The physician marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
mm
  Baseline (n=26) | 20.6 (18.7)
  Week 12 (n=26) | 11.4 (14.1)
  Week 24 (n=26) | 13.8 (14.7)
  Week 36 (n=25) | 13.1 (10.4)
  Week 48 (n=23) | 9.1 (11.3)
  Week 56 (n=25) | 13.0 (13.3)
  Week 68 (n=24) | 11.6 (11.9)
  Week 80 (n=24) | 11.3 (11.2)
  Week 92 (n=25) | 13.7 (11.7)
  Week 104 (n=25) | 10.0 (9.7)
  FU Visit 1 (n=15) | 11.7 (11.5)
  FU Visit 2 (n=25) | 15.3 (18.4)

9. Secondary Outcome: Participant's Pain Assessment Using VAS Score
Description: Participant's pain assessment was made on a horizontal 0-100 mm VAS, with 0 mm (left end of the line) described as "no pain" and 100 mm (right end of the line) as "unbearable pain". The participant marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
mm
  Baseline (n=26) | 31.9 (21.7)
  Week 12 (n=26) | 29.0 (25.1)
  Week 24 (n=26) | 33.7 (25.4)
  Week 36 (n=25) | 28.6 (21.5)
  Week 48 (n=23) | 27.8 (25.2)
  Week 56 (n=25) | 27.4 (23.1)
  Week 68 (n=24) | 27.8 (23.1)
  Week 80 (n=24) | 31.9 (24.3)
  Week 92 (n=25) | 29.5 (22.7)
  Week 104 (n=25) | 28.6 (22.6)
  FU Visit 1 (n=15) | 28.9 (25.8)
  FU Visit 2 (n=25) | 42.6 (30.1)

10. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: The Stanford HAQ-DI is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/personal care, ability to stand-up, eating, walking, hygiene, reaching, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents 'no disability' and 3 represents 'very severe, high-dependency disability'.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
units on a scale
  Baseline (n=26) | 0.68 (0.61)
  Week 12 (n=26) | 0.49 (0.43)
  Week 24 (n=26) | 0.49 (0.38)
  Week 36 (n=25) | 0.49 (0.45)
  Week 48 (n=23) | 0.48 (0.49)
  Week 56 (n=24) | 0.53 (0.60)
  Week 68 (n=24) | 0.52 (0.47)
  Week 80 (n=24) | 0.53 (0.48)
  Week 92 (n=23) | 0.43 (0.44)
  Week 104 (n=24) | 0.48 (0.50)
  FU Visit 1 (n=15) | 0.56 (0.42)
  FU Visit 2 (n=23) | 0.63 (0.59)

11. Secondary Outcome: Health Assessment Questionnaire (HAQ) Pain VAS Score
Description: The HAQ pain VAS is a measure of pain on a continuous 100 mm scale. Participants were asked to indicate how much pain they had in the past week as a result of their illness on a horizontal line from 0 (no pain) to 100 mm (severe pain).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
mm
  Baseline (n=26) | 31.9 (22.6)
  Week 12 (n=26) | 30.8 (24.5)
  Week 24 (n=26) | 37.8 (26.3)
  Week 36 (n=25) | 30.1 (23.4)
  Week 48 (n=23) | 32.7 (29.4)
  Week 56 (n=24) | 31.3 (24.0)
  Week 68 (n=24) | 32.9 (25.1)
  Week 80 (n=24) | 34.4 (27.2)
  Week 92 (n=23) | 38.2 (30.3)
  Week 104 (n=24) | 29.0 (23.9)
  FU Visit 1 (n=15) | 30.9 (24.8)
  FU Visit 2 (n=22) | 43.3 (32.8)

12. Secondary Outcome: C-Reactive Protein (CRP) Level
Description: CRP is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
milligrams per deciliter (mg/dL)
  Baseline (n=24) | 0.51 (0.91)
  Week 12 (n=26) | 3.13 (6.17)
  Week 24 (n=25) | 1.08 (1.58)
  Week 36 (n=25) | 2.58 (3.00)
  Week 48 (n=21) | 0.21 (0.27)
  Week 56 (n=24) | 0.41 (0.92)
  Week 68 (n=24) | 0.43 (0.74)
  Week 80 (n=24) | 0.64 (1.91)
  Week 92 (n=23) | 1.86 (7.11)
  Week 104 (n=25) | 0.12 (0.16)
  FU Visit 1 (n=13) | 0.10 (0.11)
  FU Visit 2 (n=24) | 1.46 (5.05)

13. Secondary Outcome: ESR Level
Description: ESR is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, and FU Visit 1 (Week 108), FU Visit 2 (Week 116)
Population: ITT population. Here, n=Number of participants analyzed for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
mm/hr
  Baseline (n=26) | 9.8 (10.2)
  Week 12 (n=24) | 4.9 (3.1)
  Week 24 (n=25) | 8.5 (7.6)
  Week 36 (n=25) | 4.6 (3.2)
  Week 48 (n=21) | 5.1 (4.7)
  Week 56 (n=24) | 4.9 (5.3)
  Week 68 (n=23) | 6.7 (7.2)
  Week 80 (n=24) | 6.4 (9.1)
  Week 92 (n=24) | 7.5 (9.2)
  Week 104 (n=25) | 5.5 (6.3)
  FU Visit 1 (n=13) | 4.8 (5.0)
  FU Visit 2 (n=24) | 21.9 (29.7)

ADVERSE EVENTS:
Time Frame: From Baseline up to approximately 2 years
Description: ITT population
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 4/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=26)
Ischaemic stroke (Nervous system disorders) | 1
Total lung capacity decreased (Investigations) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Corneal perforation (Injury, poisoning and procedural complications) | 1
Diverticulitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=26)
Chest pain (Cardiac disorders) | 2
Labyrinthitis (Ear and labyrinth disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Diarrhoea NOS (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 2
Respiratory tract infection NOS (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 7
Tonsillitis (Infections and infestations) | 4
Dengue fever (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Injury (Injury, poisoning and procedural complications) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 6
Hypercholesterolemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Osteopenia (Metabolism and nutrition disorders) | 2
Osteoporosis (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Musculoskeletal pain (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 3
Leukocyturia (Renal and urinary disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Respiratory, thoracic and mediastinal disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension NOS (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.